CLINICAL TRIAL: NCT02319798
Title: Telephone Consultation as a Substitute for Routine Out-patient Face-to-face Consultation for Children With Inflammatory Bowel Disease: Randomised Controlled Trial and Economic Evaluation.
Brief Title: Telephone Consultation as a Substitute for Routine Out-patient Face-to-face Consultation for Children With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBDV227APR2010
Record Dates: First submitted 2014-04-14; First posted 2014-12-18 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's disease; ulcerative colitis; Inflammatory bowel disease; IBD
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

ARMS (2):
- face-to-face consultations (Active Comparator): Those randomized to face-to-face follow up will attend their appointments in hospital as usual.
  Interventions: Other: face-to-face consultations
- telephone consultations (Experimental): Those randomized to telephone consultation will be told to expect a call from the gastroenterology doctor at the time of their appointment.
  Interventions: Other: telephone consultations

INTERVENTIONS:
Other: telephone consultations — Those randomized to telephone consultation will be told to expect a call from the gastroenterology doctor at the time of their appointment.
  Arms: telephone consultations
Other: face-to-face consultations — Those randomized to face-to-face follow up will attend their appointments in hospital
  Arms: face-to-face consultations

SUMMARY:
Inflammatory bowel disease (IBD) refers to two chronic diseases (Crohn's disease and ulcerative colitis) that affect the intestines. The number of new cases of IBD in people younger than 16 years old has been increasing in the United Kingdom (UK), and is currently estimated to be 700 new cases every year. There is no cure for IBD and patients experience episodes of flareups in between periods of wellbeing.

Traditionally, children with IBD are asked to attend regular hospital appointments. This means that, even if they are well, they have to get to the hospital and this can involve travelling long distances.

Telephone consultations have been shown to be beneficial in some areas of medicine but this approach has not been well studied in children. The aims of this study are to determine whether telephone consultations would improve quality of life, patient satisfaction, proportion of consultations attended and whether they would be safe and reduce costs for patients and the National Health Service (NHS). Investigators plan a randomised controlled trial involving 92 participants recruited from amongst the 250 children and adolescents aged between 8 and 16 years who attend the regional paediatric IBD centre in Manchester. Half will be assigned to telephone consultations, and half to face to face consultations. The study would have the approval of the local ethics committee and participants would have provided written consent. Investigators will compare outcomes in the two groups over 2 years. If telephone consultations prove to be effective, the NHS could offer children with IBD the choice of either telephone consultation or face to face consultation for their outpatient followup. Those who are doing well would not have to make unnecessary journeys to the hospital. This would free up clinic spaces and allow patients who are unwell, and new patients to be seen more quickly, thus reducing waiting

DETAILED DESCRIPTION:
HYPOTHESIS Telephone consultation is effective, safe, and a cost-effective alternative to traditional routine face-to-face consultation for children and adolescents with IBD.

AIMS

The specific aims of the study are:

1. To determine if telephone consultation, compared to face-to-face consultation is effective for children and adolescents with IBD.

   The investigators hypothesise that compared to face-face-consultations, telephone consultations would:
   1. improve patients' health-related quality of life
   2. have a positive impact on patient/carer satisfaction with consultations
   3. reduce out-patient non-attendance rate
2. To determine any adverse events associated with routine telephone consultations in children and adolescents with IBD.

   The investigators hypothesise that compared to face-to-face consultations, telephone consultations will not:
   1. adversely affect patients' disease course such as the number of relapses, number of hospital admissions, and number of times they have to visit their paediatrician or General Practitioner (GP) because of concerns about symptoms
   2. adversely affect the child's growth
3. To compare NHS resource utilisation, costs to the NHS and costs to patients and their carers in the two groups.

The investigators hypothesise that telephone consultations, compared to face-to-face consultations, will:

1. reduce NHS resource use
2. reduce out-patient non-attendance rate
3. be cost-effective to the NHS and
4. reduce IBD-related costs for patients and families.

METHODS SETTING AND PARTICIPANTS The study will be based at the Royal Manchester Children's Hospital, a regional Paediatric Gastroenterology referral centre. Children and adolescents with IBD from the North West of England and beyond are referred to this centre. Any patient who is aged between 8 and 16 years with a diagnosis of IBD will be eligible for entry into the trial. Eligible patients will be identified through the hospital's paediatric IBD database. There are currently about 250 eligible patients who attend the centre. Inclusion criteria are: patients aged between 8 and 16 years; diagnosis of IBD by established clinical, endoscopic, histological and radiological criteria; clinical remission defined as an abbreviated Paediatric Crohn's Disease Activity Index (aPCDAI) score of ≤10 (12) for patients with Crohn's disease or as a Paediatric Ulcerative Colitis Activity Index (PUCAI) score of <10 (13) for those with ulcerative colitis and indeterminate colitis; parental and child's consent to participate in the study. Exclusion criteria are active disease (aPCDAI>15 or PUCAI ≥15), and unwillingness to provide informed consent.

STUDY DESIGN A randomised controlled trial comparing telephone consultations with standard face-to-face out-patient consultations. It will be accompanied by an economic evaluation.

PLAN OF STUDY The investigators will send a letter of invitation to participate in the study and a research information sheet outlining the nature and importance of the study to eligible patients and their parents. The invitation letter will explicitly state that if they do not wish to take part in the study, it will not prejudice the quality of health care provision from the hospital. Two weeks later, the investigators will telephone all those who have not already responded, offering an invitation to participate and to answer any queries. Those who can not be contacted by telephone will be sent a second letter. Those who agree to take part will be interviewed by an investigator who will provide full information about the trial and obtain written informed consent. Prior to randomization, the following baseline demographic and clinical features will be recorded: patient's initials, date of birth, gender, hospital number, and disease activity (aPCDAI or PUCAI score). Participants will be provided with the contact details of relevant investigators.

Randomization

By means of a computer-generated random number, participants will be randomly allocated to one of two groups:

Intervention Group: telephone consultations Control Group: face-to-face consultations

The investigators will use a stratified block randomization with blocks of random sizes, and stratify by type of disease (i.e.Crohn's disease or ulcerative colitis/indeterminate colitis).

To ensure allocation concealment, the computer-generated assignment schedule will be held centrally and administered by 2 designated administrators who are not involved in the study. If a participant meets the inclusion criteria and provides informed consent, he or she will be entered into the study. Investigators will telephone the designated administrators, who after recording the patient's identification number, date of birth and disease activity score, will assign the next number in the series to determine allocation group. The assigned group will be recorded and implemented. Nobody will be able to alter the assignment. Participants in the telephone group will, however, retain the option to return to routine care through non-concordance with the allocated intervention.

Procedures Patients in both groups will be offered out-patient appointment dates and times. Those randomized to face-to-face follow up will attend their appointments in hospital as usual. Those randomized to telephone consultation will be told to expect a call from the gastroenterology doctor at the time of their appointment (which will be after school hours). The consulting doctor will contact the patient and parents via a telephone number (home or mobile) that the parents and patient had previously supplied as the number they would like to be contacted on. As much as possible, parents and patients will be advised to be together at the time of the appointment in order to allow both of them to participate in the consultation as is usual in practice. Up to 3 attempts within 20 minutes will be made to contact patients by phone. Details about each consultation including date and time, who was present, duration of consultations, and failed attempts at phone calls will be recorded. Patients who "DNA" an appointment in either group will be sent another appointment in accordance with normal practice.

Apart from being randomised to telephone or face-to-face consultation, routine care will be the same for patients in both groups. For instance, all patients on treatments such as azathioprine and methotrexate will continue to have relevant tests such as full blood count and liver function tests monitored regularly according to current guidelines. In our current practice, this routine monitoring does not usually take place at the routine out-patient visits but rather at the child's GP surgery, or local hospital and the results communicated to our inflammatory bowel disease nurse specialists. This practice will remain the same for all patients. It will also be emphasized that, as it is in normal practice, if a participant experiences any symptoms that cause concern at any time during the study, the parent/child should contact the IBD nurse for advice and an appropriate arrangement for assessment will be made. A relapse will not require withdrawal but the patient will be seen and treated as appropriate and will remain in the same study group.

OUTCOME MEASURES Primary outcome measure The primary outcome measure will be changes in the paediatric IBD-specific health-related quality of life (QOL) scores. QOL scores will be assessed at baseline, and 6-monthly over the 2-year follow-up period using the validated paediatric IBD QOL IMPACT questionnaire (Appendix 1). The IMPACT questionnaire was originally developed for use in paediatric IBD in Canada (14) and with minor adaptations, the questionnaire was subsequently validated in Canada ((15), the Netherlands (16), and the UK (17). The questionnaire consists of 35 questions measuring six quality of life domains (IBD symptoms, systemic symptoms, emotional functioning, social functioning, body image, and treatment/interventions) and utilizes a Likert scale to report the patient's answers. Responses are scored (from 0 to 4) and summed to give a total score (range 0 to 140). Higher scores represent better QOL.

Secondary outcome measures

1. Relapses For each participant, the number of relapses during the study period will be recorded. For patients with Crohn's disease, a relapse will be defined as an aPCDAI of >15. The PCDAI was originally developed and validated in several centres (18) and has been used widely in paediatric clinical trials. The original PCDAI includes three history items (abdominal pain, number of liquid stools, general wellbeing), five physical examination items (abdominal examination, perirectal disease, extraintestinal manifestations, weight, height velocity), and three laboratory tests (hematocrit, albumin, erythrocyte sedimentation rate). Among other things, the original PCDAI has been criticized because of the inclusion of blood tests. Recent studies have shown that an abbreviated version of the PCDAI (aPCDAI) which omits laboratory items is accurate and predicted disease activity as well as the original PCDAI (12,19). The aPCDAI consists of the three history items (abdominal pain, number of liquid stools, and general well-being), and the three physical examination items (weight loss, abdominal examination, and perirectal disease) of the original PCDAI. In order to avoid repeated blood sampling for research purposes, we will use the aPCDAI (Appendix II). Items in this index are scored on a three-point scale (zero, 5, or 10 points) and scores range from zero to 60 with higher scores indicating more active disease.

   For patients with ulcerative colitis and indeterminate colitis, a PUCAI score of >15 will be considered as a relapse. The PUCAI is a validated instrument that includes six history items (abdominal pain, rectal bleeding, stool consistency, nocturnal stools and activity level) (13). PUCAI scores can range from zero to 85 with higher scores indicating more active disease.
2. Basic anthropometric measures at every routine follow up visit / consultation Weight and height will be measured at baseline and during the routine follow up appointments in both groups. For those allocated to face to face consultations, their height and weight will be measured at their out-patients visits. For children allocated to telephone consultations, height and weight will be measured by their local paediatric service, prior to their telephone appointment. A member of the study team will, prior to each follow up period, contact those in the telephone consultation group to remind them to the have measurements done. A study team member will then contact the local service or the parent / patient to obtain the measurements. Height and body mass index (BMI) z scores will be calculated based on sex- and age-related UK centile charts.
3. Patient satisfaction with consultations - to be completed after every Participants or their carers will be asked to complete a Consultation Satisfaction Questionnaire (CSQ) at the end of each consultation. This CSQ is an 18 item consultation-specific satisfaction measure that was developed and validated by Baker (20, 21). It has since been used in other areas/settings including community nursing (22, 23), and has recently been modified and tested for use in consultations involving patients aged 15 years or younger (24). After discussions with the originator of this instrument and the researcher who modified it for paediatric use, the modified version of the CSQ will be adapted for children aged 15 years and younger (Appendix IIa), and the original version adapted for patients aged 16 years or older (Appendix IIb) {R Baker and P Kinnersley, personal communication, July 2008}.
4. Number of hospital admissions for IBD over 24 months. Data will be obtained from the patient's hospital records.
5. Proportion of out-patient consultations attended For each group, the proportion of outpatient appointments attended over the 24-month follow-up period will be calculated by dividing the total number of appointments (telephone or face-to-face) offered by the number of appointments attended.
6. Duration of consultations The duration of each consultation will be recorded in the patient's medical notes.
7. Adverse effects of immuno-suppressive agents such as azathioprine and methotrexate.

   Any adverse effect of immuno-suppressive agents that participants may be receiving during the study period will be recorded.
8. Economic evaluation Investigators will assess the use of health care resources, costs to the NHS and costs to patients and their carers in the two groups. Data on resource use in tertiary, secondary and primary care will be collected. Data on resources used for outpatient consultations (telephone or face-to-face), additional or unscheduled hospital visits, tests and procedures, drug prescriptions, hospital admissions, and general practice visits will be identified for every patient.

At each outpatient consultation (telephone or face-to-face), the clinician will record details of the consultation including date of the visit and duration of the consultation. Abortive telephone calls will be recorded as well as face-to-face appointments missed. For telephone consultations, it will be noted whether calls were local, national, or made to mobile phones. Data on inpatient admissions, any investigations or procedures, and treatments received will be abstracted from the patient's hospital records. A patient/carer diary (Appendix IV) will be used to collect information on drug utilisation (name, dose, frequency, and duration), GP visits, and care received at other hospitals. Patients will be asked to complete the diary every time they visited their GP, changed their regular medications, or were seen at other hospitals. Diary information will be collated 6-monthly. Resource use that was clearly unrelated to IBD will be excluded from the economic evaluation.

Note:Routine follow ups / consultations vary between patients depending on how well they are. Patients may also be seen for routine appointments in between the scheduled study follow ups.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 8 and 16 years
* diagnosis of IBD by established clinical, endoscopic, histological and radiological criteria
* clinical remission defined as an abbreviated Paediatric Crohn's Disease Activity Index (aPCDAI) score of ≤10 for patients with Crohn's disease or as a Paediatric Ulcerative Colitis Activity Index (PUCAI) score of <10 for those with ulcerative colitis and indeterminate colitis
* parental and child's consent to participate in the study.

Exclusion Criteria:

* active disease (aPCDAI>15 or PUCAI ≥15)
* unwillingness to provide informed consent.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in the paediatric IBD-specific health-related quality of life (QOL) scores. | 6 monthly over 2 years
  QOL scores will be assessed at baseline, and 6-monthly over the 2-year follow-up period using the validated paediatric IBD QOL IMPACT questionnaire

SECONDARY OUTCOMES:
Relapses | All relapses over 2 years
  For each participant, the number of relapses during the study period will be recorded. For patients with Crohn's disease, a relapse will be defined as an aPCDAI of >15. The aPCDAI consists of the three history items (abdominal pain, number of liquid stools, and general well-being), and the three physical examination items (weight loss, abdominal examination, and perirectal disease). Items in this index are scored on a three-point scale (zero, 5, or 10 points) and scores range from zero to 60 with higher scores indicating more active disease.
  For patients with ulcerative colitis and indeterminate colitis, a PUCAI score of >15 will be considered as a relapse. The PUCAI is a validated instrument that includes six history items (abdominal pain, rectal bleeding, stool consistency, nocturnal stools and activity level). PUCAI scores can range from zero to 85 with higher scores indicating more active disease.

OTHER OUTCOMES:
Patient satisfaction with consultations | every appointment during study period ( over 2 years)
  Participants or their carers will be asked to complete a Consultation Satisfaction Questionnaire (CSQ) at the end of each consultation. This CSQ is an 18 item consultation-specific satisfaction measure that was developed and validated by R Baker (Br J Gen Pract 1990;40:487-90. and Dialogue, 3rd edition. Clinical Governance Research and Development Unit, University of Leicester. 2001)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Manchester Children's Hospital, Manchester, Lancs, United Kingdom

REFERENCES:
- [Derived] Akobeng AK, O'Leary N, Vail A, Brown N, Widiatmoko D, Fagbemi A, Thomas AG. Telephone Consultation as a Substitute for Routine Out-patient Face-to-face Consultation for Children With Inflammatory Bowel Disease: Randomised Controlled Trial and Economic Evaluation. EBioMedicine. 2015 Aug 8;2(9):1251-6. doi: 10.1016/j.ebiom.2015.08.011. eCollection 2015 Sep. PMID 26501125